CLINICAL TRIAL: NCT04552535
Title: Real-World Effectiveness of Afatinib (Gilotrif) Following Immunotherapy in the Treatment of Metastatic, Squamous Cell Carcinoma of the Lung: A Multi-Site Retrospective Chart Review Study in the U.S.
Brief Title: A Study in the United States Using Electronic Medical Records (EMR) to Assess Effectiveness of Afatinib (Gilotrif) Following Pembrolizumab and Chemotherapy in the Treatment of Metastatic Squamous Cell Carcinoma of the Lung
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200-0325
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Second line (2L) afatinib: Second line (2L) afatinib treated following discontinuation of pembrolizumab in combination with platinum-based doublet chemotherapy (first line (1L))
  Interventions: Drug: Second line (2L) afatinib
- Second line (2L) chemotherapy: Second line (2L) chemotherapy treated following discontinuation of pembrolizumab in combination with platinum-based doublet chemotherapy (first line (1L))
  Interventions: Drug: Second line chemotherapy

INTERVENTIONS:
Drug: Second line (2L) afatinib — Afatinib
  Groups: Second line (2L) afatinib
Drug: Second line chemotherapy — Chemotherapy
  Groups: Second line (2L) chemotherapy

SUMMARY:
This study aims to characterize the profile and outcomes for patients with Squamous Cell Carcinoma of the Lung (SqCC) who progress on 1L pembrolizumab in combination with platinum based chemotherapy and receive afatinib as second line (2L) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of squamous or mixed histology non-small cell lung cancer
* Treated with pembrolizumab in combination with platinum-based chemotherapy as initial therapy for advanced or metastatic disease (stage IIIB or IV)

  * First cycle of pembrolizumab received after 06/01/2018
  * Permanently discontinued 1L pembrolizumab treatment
* Initiated second-line treatment at least 3 months prior to the date of data collection, with either :

  * Afatinib
  * Any chemotherapy
* Age ≥ 18 years

Exclusion Criteria:

-Received pembrolizumab in combination with platinum-based chemotherapy as part of an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic Squamous cell carcinoma (SqCC) of the lung treated with pembrolizumab in combination with platinum doublet chemotherapy as first line (1L) treatment followed by either afatinib as second line (2L) treatment or chemotherapy as 2L treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardinal Health Specialty Solutions, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This retrospective, non-interventional, multi-site cohort study utilized existing data from the electronic medical records of patients with advanced or metastatic Squamous Cell Carcinoma (SqCC) of the lung treated with first-line pembrolizumab in combination with platinum-doublet chemotherapy, followed by second-line afatinib or chemotherapy.
Pre-assignment Details: All patients (pts) aged ≥18 years, initiated first-line (1L) pembrolizumab and platinum-based combination chemotherapy (CT) after 1st June 2018, and subsequently discontinued 1L therapy. All pts had started second-line treatment with either afatinib or any CT at least 3 months prior to date of data collection. Maximum follow-up for any pts was approx 15 months. Pts were excluded if they had received pembrolizumab in combination with platinum-based CT as part of an interventional clinical trial.
Groups:
- Second-line Afatinib Treatment Group: Patients in the second-line afatinib treatment group initiated first-line pembrolizumab and platinum-based combination chemotherapy after 1st June 2018, and subsequently discontinued first-line therapy. All patients had started second-line treatment with afatinib at least 3 months prior to the date of data collection.
- Second-line Chemotherapy Treatment Group: Patients in the second-line chemotherapy treatment group initiated first-line pembrolizumab and platinum-based combination chemotherapy after 1st June 2018, and subsequently discontinued first-line therapy. All patients had started second-line treatment with any chemotherapy at least 3 months prior to the date of data collection.
Period: Overall Study
Arm/Group | Second-line Afatinib Treatment Group | Second-line Chemotherapy Treatment Group
Started | 99 | 101
Completed | 99 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients (pts) aged ≥18 years, initiated first-line (1L) pembrolizumab and platinum-based combination chemotherapy (CT) after 1st June 2018, and subsequently discontinued 1L therapy. All pts had started second-line treatment with either afatinib or any CT at least 3 months prior to date of data collection. Maximum follow-up for any pts was approx 15 months. Pts were excluded if they had received pembrolizumab in combination with platinum-based CT as part of an interventional clinical trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Second-line Afatinib Treatment Group | Second-line Chemotherapy Treatment Group | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 67 [60 to 71] | 66 [61 to 70] | 67 [61 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 34 | 77
  Male | 56 | 67 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 23 | 53
  White | 59 | 73 | 132
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Tumor histology [Count of Participants; unit: Participants]
  Squamous cell only | 64 | 98 | 162
  Mixed histology | 35 | 3 | 38
Epidermal growth factor receptor (EGFR) mutation status [Count of Participants; unit: Participants]
  EGFR mutation positive | 39 | 5 | 44
  EGFR mutation negative | 28 | 33 | 61
  Not tested / unknown | 32 | 63 | 95
Smoking history [Count of Participants; unit: Participants]
  Never smoked | 12 | 0 | 12
  Current smoker | 16 | 19 | 35
  Former smoker | 71 | 82 | 153
Eastern Cooperative Oncology Group Performance Status at initiation of second line (2L) treatment [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status (ECOG PS) is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    ECOG 0/1 | 45 | 50 | 95
    ECOG ≥ 2 | 54 | 51 | 105
Tumor stage at initial diagnosis [Count of Participants; unit: Participants] — Disease stage means how big tumor is + how far it has spread. They range from 0 (not spread) to IV (spread throughout body). 0 - cancer not spread beyond inner lining of affected organ; I - is small and not spread to lymph nodes (LN); II - spread to some LN near original tumor; III - spread to nearby tissue or spread to far away LN (IIIA: heterogeneous group with diversity of tumor characteristics and varying degrees of LN involvement; IIIB: involves LN on opposite side of chest or above collar bone, or heart or trachea + LN in chest center or near windpipe); IV - has spread to other organs.
  Participants
    Tumor stage I to IIIA | 13 | 8 | 21
    Tumor stage IIIB | 7 | 3 | 10
    Tumor stage IV | 79 | 90 | 169
Sites of metastatic disease at initiation of second line treatment [Count of Participants; unit: Participants]
  Liver | 65 | 69 | 134
  Contralateral lung nodule | 51 | 43 | 94
  Blood and bone marrow | 41 | 47 | 88
  Adrenal gland | 26 | 48 | 74
  Pleura (nodules, effusion) | 24 | 21 | 45
  Intra-abdominal lymph nodes | 19 | 14 | 33
  Brain | 14 | 10 | 24
Most common comorbidities at initiation of second line treatment [Count of Participants; unit: Participants]
  Any comorbidity | 98 | 88 | 186
  Hypertension | 62 | 56 | 118
  Chronic pulmonary disease | 35 | 49 | 84
  Cardiovascular disease | 23 | 33 | 56
  Depression | 27 | 14 | 41
  Diabetes without chronic complications | 21 | 16 | 37
Radiation therapy [Count of Participants; unit: Participants]
  First line or prior | 14 | 10 | 24
  Second line | 12 | 9 | 21
Programmed death ligand 1 (PD-L1) expression level [Count of Participants; unit: Participants]
  <1% | 26 | 30 | 56
  1 to 49% | 55 | 54 | 109
  >50% | 15 | 6 | 21
  Not tested | 3 | 11 | 14

OUTCOME MEASURES:

1. Primary Outcome: Time on Treatment With Afatinib or Chemotherapy During Second Line (2L) Treatment
Description: Time on treatment was defined as the interval from the start of second-line treatment until discontinuation of second-line treatment for any reason, e.g. toxicity, progression, death, patient choice. The end of 2L treatment was defined as the date of last treatment order for afatinib plus the days of supply on the last known treatment order up to the date of data collection (but not exceeding). The Kaplan-Meier (KM) method was used to estimate the median and 95% confidence interval for time on treatment.
Time Frame: From the start of second-line treatment until discontinuation of second-line treatment, up to 12.3 months for afatinib treated and up to 7.5 months for chemotherapy treated patients
Population: All patients (pts) who initiated first-line (1L) pembrolizumab and platinum-based combination chemotherapy (CT) after 1st June 2018, and subsequently discontinued 1L therapy and had started second-line treatment with either afatinib or any CT at least 3 months prior to date of data collection.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Second-line Afatinib Treatment Group | Second-line Chemotherapy Treatment Group
Number analyzed (Participants) | 99 | 101
months | 7.3 [5.2 to 8.1] | 4.2 [3.9 to 4.9]

2. Primary Outcome: Time on Treatment With Afatinib During Second Line (2L) Treatment Defined by Histology Status
Description: Time on treatment was defined as the interval from the start of second-line treatment until discontinuation of second-line treatment for any reason, e.g. toxicity, progression, death, patient choice. The end of 2L treatment was defined as the date of last treatment order for afatinib plus the days of supply on the last known treatment order up to the date of data collection (but not exceeding). The Kaplan-Meier (KM) method was used to estimate the median and 95% confidence interval for time on treatment. Patients treated with afatinib were analysed for their histology status and categorized into a squamous cell - or mixed histology treatment group.
Time Frame: From the start of second-line treatment until discontinuation of second-line treatment, up to 12.3 months for afatinib treated patients
Population: All patients (pts) who initiated first-line (1L) pembrolizumab and platinum-based combination chemotherapy (CT) after 1st June 2018, and subsequently discontinued 1L therapy and had started second-line treatment with afatinib at least 3 months prior to date of data collection. Only patients treated with afatinib and with squamous cell - or mixed histology were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Second-line Afatinib Treatment Group With Squamous Cell Histology: Patients in the second-line afatinib treatment group with squamous cell histology initiated first-line pembrolizumab and platinum-based combination chemotherapy after 1st June 2018, and subsequently discontinued first-line therapy. All patients with squamous cell histology had started second-line treatment with afatinib at least 3 months prior to the date of data collection.
- Second-line Afatinib Treatment Group With Mixed Histology: Patients in the second-line afatinib treatment group with mixed histology initiated first-line pembrolizumab and platinum-based combination chemotherapy after 1st June 2018, and subsequently discontinued first-line therapy. All patients with mixed histology had started second-line treatment with afatinib at least 3 months prior to the date of data collection.
Arm/Group | Second-line Afatinib Treatment Group With Squamous Cell Histology | Second-line Afatinib Treatment Group With Mixed Histology
Number analyzed (Participants) | 64 | 35
months | 5.8 [4.4 to 8.0] | 8.1 [5.5 to 9.9]

3. Primary Outcome: Time on Treatment With Afatinib During Second Line (2L) Treatment Defined by Epidermal Growth Factor Receptor (EGFR) Mutation Status
Description: as for outcome 1
Time Frame: as for outcome 2
Population: All patients (pts) who initiated first-line (1L) pembrolizumab and platinum-based combination chemotherapy (CT) after 1st June 2018, and subsequently discontinued 1L therapy and had started second-line treatment with afatinib at least 3 months prior to date of data collection. Only afatinib treated patients with an EGFR mutation positive or negative status were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Second-line Afatinib Treatment Group With Epidermal Growth Factor Receptor Mutation Positive Status: Patients in the second-line afatinib treatment group with EGFR mutation positive status initiated first-line pembrolizumab and platinum-based combination chemotherapy after 1st June 2018, and subsequently discontinued first-line therapy. All patients with EGFR mutation positive status had started second-line treatment with afatinib at least 3 months prior to the date of data collection.
- Second-line Afatinib Treatment Group With Epidermal Growth Factor Receptor Mutation Negative Status: Patients in the second-line afatinib treatment group with Epidermal growth factor receptor (EGFR) mutation negative status initiated first-line pembrolizumab and platinum-based combination chemotherapy after 1st June 2018, and subsequently discontinued first-line therapy. All patients with EGFR mutation negative status had started second-line treatment with afatinib at least 3 months prior to the date of data collection.
Arm/Group | Second-line Afatinib Treatment Group With Epidermal Growth Factor Receptor Mutation Positive Status | Second-line Afatinib Treatment Group With Epidermal Growth Factor Receptor Mutation Negative Status
Number analyzed (Participants) | 39 | 28
months | 7.4 [5.6 to 8.6] | 5.9 [4.4 to NA] — not estimable due to unsufficient events

4. Primary Outcome: Number of Patients With Severe Immune-related Adverse Events (irAEs) of Specific Interest During Second-line Treatment
Description: Chart abstractors (i.e. the patients treating physician) were asked to abstract information regarding severe (grade 3 or higher) irAEs of specific interest (including pneumonitis, colitis, hepatitis, interstitial lung disease, higher indeterminate pulmonary events, death, or discontinuation of therapy due to toxicity) during first line (1L) treatment and second line (2L) for both patients treated with afatinib in 2L and those treated with chemotherapy in 2L. Providers/abstractors were asked only if these specific immune related events occurred.
Time Frame: From the start of second-line treatment to the end of follow-up, up to 15 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Second-line Afatinib Treatment Group | Second-line Chemotherapy Treatment Group
Number analyzed (Participants) | 99 | 101
Participants | 6 | 0

ADVERSE EVENTS:
Time Frame: From the start of second-line treatment to the end of follow-up, up to 15 months.
Description: Adverse events (AEs) were only collected and reported for 2L afatinib treatment group according to protocol requirements.
  All 2L afatinib treatment group patients (pts) who initiated first-line (1L) pembrolizumab and platinum-based combination chemotherapy (CT) after 1st June 2018, and subsequently discontinued 1L therapy and had started second-line (2L) treatment with afatinib at least 3 months prior to date of data collection.
  Serious AEs were not collected and reported for this study.
Arm/Group | Second-line Afatinib Treatment Group
All-Cause Mortality (participants affected / at risk) | 2/99
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 37/99
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Second-line Afatinib Treatment Group (N=99)
Diarrhea (Gastrointestinal disorders) | 26
Skin rash (Skin and subcutaneous tissue disorders) | 6
Fatigue (General disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT04552535/Prot_SAP_000.pdf